CLINICAL TRIAL: NCT00913172
Title: Improving Community Based TB Care in Southern Ethiopia Cost and Cost Effectiveness
Brief Title: Cost and Cost-effectiveness of PTB+ Treatment in Southern Ethiopia
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Responsible Party: Bernt Lindtjørn, Professor, University of Bergen
Other Study IDs: 000001
Record Dates: First submitted 2009-05-28; First posted 2009-06-04 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2009-05

CONDITIONS: Smear-positive TB Cases
Keywords: TB; cost; HEWs; Cost-effectiveness; treatment success rate
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group: Directly Observed Treatment under Health Extension Workers
  Interventions: Other: Treatment
- Control group: Directly observed treatment under general health workers

INTERVENTIONS:
Other: Treatment — Directly observed treatment (DOT) by health extension workers (HEWs)
  Other Names: community based TB care
  Groups: Intervention group

SUMMARY:
Evidences for policy making and decision related to the cost of delivering tuberculosis (TB) control is lacking in Ethiopia. The investigators aimed to determine the cost and cost-effectiveness of involving health extension workers (HEWs) in TB treatment under the community-based initiative in Ethiopia.

DETAILED DESCRIPTION:
Two treatment options were compared - health facility and community DOT. In 1995, Ethiopia adopted World Health Organization (WHO) recommended DOTS strategy for TB control. The treatment regimen for new smear-positive patients includes two months of ethambutol, rifampicin, isoniazid and pyrazinamide followed by six months of ethambutol and isoniazid. For children the continuation phase treatment was replaced by four months of rifampicin and isoniazid. Follow up sputum examinations were conducted at the end of 2, 5 and 7 months treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary tuberculosis suspects of any age and sex

Exclusion Criteria:

* Healthy individuals or non tuberculosis patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted along a CRT to find out if involving HEWs improves the treatment success rate of smear-positive patients. For both treatment alternatives, smear-positive patients who were diagnosed (from September 2006 to September 2007) and started treatment were prospectively enrolled until the end of treatment. The detail of the study are given elsewhere
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
cost per successfully treated smear-positive case | September 2006 to April 2008

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Datiko, MD, Principal Investigator — UoB, RHB; Bernt Lindtjorn, MD, PhD, Study Director — UoB
Locations (1):
- YAHC, Irgalem, Snnpr, Ethiopia

REFERENCES:
- [Result] Datiko DG, Lindtjorn B. Cost and cost-effectiveness of smear-positive tuberculosis treatment by Health Extension Workers in Southern Ethiopia: a community randomized trial. PLoS One. 2010 Feb 17;5(2):e9158. doi: 10.1371/journal.pone.0009158. PMID 20174642